CLINICAL TRIAL: NCT04347460
Title: Establishing a Covid-19 Prospective Cohort to Document Cases of Secondary Hemophagocytic Lymphohistiocytosis (sHLH, Synonoums to Macrophage Activation Syndrome)
Brief Title: Establishing a COVID-19 Prospective Cohort for Identification of Secondary HLH
Acronym: COVIDHLH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 161/20 S
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: COVID
Keywords: MAS; HLH; COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID 19: Patients requiring ICU treatment due to severe COVID 19 interstitial pneumonia or otherwise COVID-19 related disease

SUMMARY:
SARS-CoV2 has become a pandemic disease putting an enormous burden on health care systems around the world. A considerable amount of patients require intensive care treatment for Covid-19 associated pneumonia. At this point there is no specific treatment, apart from supportive intensive care treatment protocols for severe COVID-19 disease.The latest reports describe massive hyperinflammation in some of the severe COVID-19 patients, which is not a typical finding in virus associated pneumonia. The H-score and the modified HLH 2004 score offer diagnostic tools, that help establishing the diagnosis of HLH. Even more important is the expert clinical judgment to establish the diagnosis of sHLH.

DETAILED DESCRIPTION:
SARS-CoV2 has become a pandemic disease putting an enormous burden on health care systems around the world. The course of disease is relatively mild in most of the patients, but there is a considerable amount of patients that require intensive care treatment for Covid-19 associated pneumonia. At this point there is no specific treatment, apart from supportive intensive care treatment protocols for severe COVID-19 disease.The latest reports describe massive hyperinflammation in some of the severe COVID-19 patients. The H-score and the modified HLH 2004 score offer diagnostic tools, that helps establishing the diagnosis of HLH. Moreover expert clinical judgment is key to establish a diagnosis of sHLH. Still, so far no systematic analysis has been carried out answering the question as to whether or not these patients suffer from secondary HLH and could potentially benefit from immunomodulatory drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17a
* diagnosis of SARS CoV 2 by PCR testing
* Hospitalized due to clinical severity of the disease
* written and informed consent or consent of the family
* GFR<30 is not an exclusion criterion

Exclusion Criteria:

* not fulfilling the inclusion criteria
* missing written and informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will recruit patients with COVID 19 interstital pneumonia with need of ICU treatment at the Klinikum rechts der Isar.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Presence of sHLH as determined by expert chart review by two independent reviewers | in the first week after admission to the ICU
  blinded chart review by a hematooncologist and a rheumatologist having expert experience in HLH diagnosis and treatment
Determine the incidence of patients fulfilling HLH criteria in Covid 19 viral infection | in the first week after admission to the ICU
  Calculate HScore in all recruited patients
Determine the incidence of patients fulfilling modified 2004 HLH diagnostic criteria (Ferritin > 10000 μg/L) in Covid 19 viral infection | in the week after admission to the ICU
  Calculate modified 2004 HLH diagnostic criteria in all study participants
Characterization and incidence of the hyper-inflammatory state in COVID-19 | assessed within 15 days post ICU-admission
  characterized by sIL-2, Ferritin, Il-6, CRP, PCT and aberrant cellular activation (differential blood count and immunophenotypic analysis)

SECONDARY OUTCOMES:
all cause mortality assesed on day 15 | assesed on study day 15
  vital status of patients will be assesed by clinical records or phone calls to patient or relatives or other hospitals involved in the care of the patient
all cause mortality assesed on day 29 | assesed on study day 29
  vital status of patients will be assesed by clinical records or phone calls to patients or relatives or other hospitals involved in the care of the patient
immunophenotpye | in the first days after admission to the ICU
  characterize immune cell populations

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schmaderer, M.D., Principal Investigator — Department of Nephrology, TUM Medical School, Klinikum rechts der Isar
Locations (1):
- Department of nephrology, Klinikum rechts der Isar, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No